CLINICAL TRIAL: NCT02284048
Title: Effect of Ticagrelor on Adenosine-Induced Coronary Flow Reserve in Patients With Microvascular Angina
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Daoquan Peng, Professor, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ISSBRIL0217
Record Dates: First submitted 2014-11-02; First posted 2014-11-05 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Microvascular Angina
Keywords: Ticagrelor; Coronary Flow Reserve
MeSH Terms: conditions — Microvascular Angina | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Placebo Comparator): nitrate,beta blocker
  Interventions: Drug: ticagrelor
- ticagrelor (Active Comparator): ticagrelor 90mg qd
  Interventions: Drug: ticagrelor

INTERVENTIONS:
Drug: ticagrelor — compare the effect of ticagrelor and control on the Coronary Flow Reserve in patients with microvessel angian
  Other Names: Brilinta

SUMMARY:
This study is undertaken to determine if ticagrelor augments adenosine-induced coronary flow reserve (CFR), ameliorates clinical symptomatology and exercise tolerance in patients with MVA

DETAILED DESCRIPTION:
Considering the reduced CFR and increased platelet aggregability in patients with MVA, together with the augmented effect on adenosine-mediated coronary blood flow and potent antiplatelet effect of ticagrelor, we speculate that ticagrelor can promisingly ameliorate the coronary microvascular function in patients with MVA.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study subjects should fulfill the following criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female or male aged 18-80 years
3. A diagnosis of stable primary MVA based on the presence of

   * a history of typical effort angina,
   * exercise-induced ST-segment depression>1 mm,
   * normal or near-normal (coronary artery stenosis<50%) coronary angiography,
   * absence vasospastic angina
   * a coronary flow reserve (CFR) <2.5 in the left anterior descending coronary artery as assessed by coronary blood flow (CBF) response to adenosine at transthoracic Doppler echocardiography
   * suboptimal control of symptoms on conventional anti-ischemic therapy, as indicated by the occurrence of >1 episode per week of angina

Exclusion Criteria:

ubjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. concomitance with any of the cardiac condition below

   * significant （>50%）coronary plaque disease
   * coronary artery spasm at angiography or other evidence of vasospastic angina
   * valvular or other structural heart disease
   * uncontrolled hypertension
   * abnormal echocardiographic examination including left ventricular hypertrophy
2. no previous consumption of the ticagrelor
3. no apparent contraindications to ticagrelor administration.

   * History of Intracranial Hemorrhage
   * Active Bleeding
   * Severe Hepatic Impairment: AST and ALT are greater than 3 times of the upper limit. Bilirubin is greater than the upper limit.
   * hypersensitivity (e.g. angioedema) to ticagrelor or any component of the product
   * severe COPD or asthma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
adenosine-induced coronary flow reserve (CFR) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Daoquan Peng, MD, PhD, Study Chair — Second Xiangya Hospital of Central South University